CLINICAL TRIAL: NCT02161198
Title: A Single-center, Randomized, Placebo-controlled, Double-blind Clinical Trial to Evaluate the Efficacy and Safety After 14-week of Ginseng Polysaccharide Extract
Brief Title: Efficacy and Safety Study of Ginseng Polysaccharide Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Health Biomed Inc. (Industry)
Responsible Party: Principal Investigator, Kyung-Soo Kim, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-75
Record Dates: First submitted 2014-06-01; First posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Panax ginseng CA; ginsan; polysaccharide; immunity; natural killer cell
MeSH Terms: interventions — ginsan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Y-75 (Experimental): volunteers receive 3 packages twice a day up to 14 weeks
  Interventions: Dietary Supplement: Y-75
- Placebo (Placebo Comparator): volunteers receive 3 packages twice a day up to 14 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Y-75 — Y-75 (1 g) and starch (1 g) as a diluting agent and were packed to contain 2 g/package
  Other Names: Ginsan
  Arms: Y-75
Dietary Supplement: Placebo — Caramel syrup (0.03 g) and starch (1.97 g) were packed identically to the active treatment
  Arms: Placebo

SUMMARY:
Y-75/ginsan is an acidic polysaccharide with a molecular weight of 150,000 Da, isolated from the aqueous Korean Panax ginseng extract. Preclinical laboratory studies have shown its function as an immunomodulatory molecule. The present study performed to evaluate the safety and beneficial effects of Y-75 on immune function in a group of healthy adults.

The focus of this trial was modulation of innate immunity, comprising cytotoxic activity of natural killer cells, phagocytic activity of polymorphonuclear leukocytes and mononuclear phagocytes, and serum levels of monocyte-derived mediators.

ELIGIBILITY:
Inclusion Criteria:

* Good general health

Exclusion Criteria:

* human immunodeficiency virus-1 infection
* malignancy
* active cardiovascular, renal, pulmonary, hepatic, neurological, psychiatric disease
* recent (within 4 weeks) acute respiratory tract symptoms
* immunosuppressive therapy including cytotoxic agents and corticosteroids
* medication (within 4 weeks) deemed likely to interfere with the evaluation
* history of allergic or other adverse reactions to ginseng products

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in natural killer cell activity from a baseline level | baseline (prior to the initial dose) , week 8, and week 14

SECONDARY OUTCOMES:
Changes from baseline in phagocytic activity of macrophages and polymorphonuclear cells | baseline, week 8, and week 14
Changes from baseline in serum levels of tumor necrosis factor-alpha and interleukin-12 | baseline, week 8, and week 14
Number of patients with laboratory abnormalities | baseline, week 8, and week 14
  Laboratory measurements included blood chemistry (BC), complete blood count (CBC), and urinalysis
Number of participants with serious and non-serious adverse events | Up to 14 weeks
  Any change from the baseline status was defined as an adverse event
Number of patients with abnormal findings in physical examination and vital signs | baseline, week 8, and week 14
  Physical examination includes body weight, ocular inspection, and heart and lung auscultation.
  Vital signs include blood pressure, heart rate, and body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Soo Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

REFERENCES:
- [Derived] Cho YJ, Son HJ, Kim KS. A 14-week randomized, placebo-controlled, double-blind clinical trial to evaluate the efficacy and safety of ginseng polysaccharide (Y-75). J Transl Med. 2014 Oct 9;12:283. doi: 10.1186/s12967-014-0283-1. PMID 25297058